CLINICAL TRIAL: NCT06698614
Title: Manganese-Enhanced Magnetic Resonance Imaging (MEMRI) in Patients With Kidney Disease
Brief Title: MEMRI and Kidney Disease
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 23/WA/0276
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury; Kidney Transplant; Vasculitis; Chronic Kidney Disease(CKD)
Keywords: manganese enhanced magnetic resonance imaging; kidney disease; MEMRI; Manganese enhanced MRI
MeSH Terms: conditions — Acute Kidney Injury; Vasculitis; Renal Insufficiency, Chronic; Kidney Diseases | interventions — Hematologic Tests; Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bloods tests- FBC, renal function, liver function.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Acute Kidney Injury: 20 patients with acute kidney injury (AKI). AKI diagnosis will be based on clinical and biochemical data reflecting KDIGO criteria.
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Blood tests; Diagnostic Test: Urine tests; Diagnostic Test: Cardiovascular analysis
- Chronic Kidney Disease: 20 age- and sex-matched patients with CKD will be recruited and the patients' eGFR will be matched to that of patients who had AKI and developed persistent renal impairment at the time of their interval scan (3-6 months from their baseline scan).
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Blood tests; Diagnostic Test: Urine tests; Diagnostic Test: Cardiovascular analysis
- Control Subjects: 20 age-, sex- and cardiovascular risk factor- matched control subjects will be recruited and matched to the AKI cohort
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Blood tests; Diagnostic Test: Urine tests; Diagnostic Test: Cardiovascular analysis
- Vasculitis: 20 patients with a new diagnosis of vasculitis (or an existing diagnosis with relapsing disease), and kidney involvement
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Blood tests; Diagnostic Test: Urine tests; Diagnostic Test: Cardiovascular analysis
- Kidney failure undergoing transplantation: 20 patients with kidney failure and will receive a kidney transplant in 1 month
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Blood tests; Diagnostic Test: Urine tests; Diagnostic Test: Cardiovascular analysis
- Kidney transplant rejection: 20 patients with a biopsy proven diagnosis of transplant rejection
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Blood tests; Diagnostic Test: Urine tests; Diagnostic Test: Cardiovascular analysis

INTERVENTIONS:
Diagnostic Test: MRI — MRI imaging of the kidney and heart with an intravenous infusion of manganese dipyridoxl diphosphate (Mangafodipir, MnDPDP).
Diagnostic Test: Blood tests — full blood count, urea and electrolytes, liver function test, CRP, biomarkers for endothelial function, storage of serum and plasma for future analyses.
Diagnostic Test: Urine tests — Urine protein, Urine creatinine
Diagnostic Test: Cardiovascular analysis — 24 hour blood pressure, arterial stiffness

SUMMARY:
Acute kidney injury (AKI) is common and costly.1 Although patients who suffer an episode of AKI may recover, many will go on to develop cardiovascular disease and chronic kidney disease (CKD). Cardiovascular disease is an important complication of AKI.2 Similar to AKI, CKD and kidney transplantation and kidney donation associations with cardiovascular disease.1 The risk of cardiovascular disease complications is also increased in patients with inflammatory diseases that affect the kidneys, such as vasculitis.

Currently, there are no reliable biomarkers that will identify those patients with kidney disease that will go on to develop cardiovascular disease. This study will explore the potential of manganese-enhanced magnetic resonance imaging (MEMRI) to act as a biomarker of AKI and its cardiovascular and renal complications. An analogue of calcium, manganese is readily taken-up into viable cells where it increases T1 relaxivity. Preliminary data show rapid manganese uptake in the heart and kidneys of healthy subjects.

The investigators propose to use MEMRI to demonstrate differences in renal and myocardial calcium handling in patients with acute insults (such as AKI, transplant rejection, donation or episodes of rejection or new vasculitis presentations) or improvements (such as transplantation). The investigators will also investigate whether these abnormalities reverse in those whose injury resolves or persist in those who clearly develop CKD, or who are at risk of future cardiovascular disease and CKD.

ELIGIBILITY:
Inclusion Criteria:

All subjects to be entered must:

Be able to provide written informed consent after having received oral and written information about the study.

>18 years of age Availability to complete study visits If female, be non-pregnant as evidenced by a negative pregnancy test or be post-menopausal or surgically sterile.

Additionally, cohort specific inclusion criteria are as follows:

Cohort 1; Acute kidney injury-

A diagnosis of AKI will be made based on the following criteria (based on the definition used in the Kidney Precision Medicine Project www.kpmp.org):

Previous (within 3 years) eGFR >45 ml/min/1.73m2 OR no history of kidney disease if no blood results available AND Elevated creatinine >1.5x previous result OR >150 μmol/L if no previous value AND Increasing creatinine within 48 hours OR requirement for dialysis.

Cohort 2; Chronic kidney disease- Stable CKD for at least 6 months (monitored by eGFR), matched to AKI cohort at follow up based on renal function.

Cohort 3: Matched controls- Matched to AKI cohort participants at baseline for age, sex, cardiovascular disease risk and cardiovascular medication.

Cohort 4; Vasculitis- A new diagnosis of vasculitis or an existing diagnosis with relapsing disease, and kidney involvement.

Cohort 5; Kidney transplantation- Has kidney failure and has received a kidney transplant in the preceding 1 month.

Cohort 6: Kidney transplant rejection- Biopsy proven episode of transplant rejection.

Exclusion Criteria:

The following criteria apply to all patients:

1. Unable to give informed consent.
2. Have any contraindications to standard MRI safety criteria, including implanted devices.
3. Subjects under the age of 18 years old.
4. Pregnancy/positive pregnancy test.
5. Current breastfeeding.
6. Have a diagnosis of kidney disease due to polycystic kidney disease.
7. Patients in critical care or on surgical wards will be excluded.
8. Patients taking calcium channel antagonists or digoxin.

Additionally, cohort specific exclusion criteria are as follow:

Cohort 1- Excluded if they have a diagnosis of diabetes. Cohort 2- Excluded if receiving dialysis or those with a functional kidney transplant, multi-system disorders (e.g., systemic vasculitis), or any patients receiving immunosuppression.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cohort 1- Acute Kidney Injury- 20 patients with acute kidney injury (AKI). AKI diagnosis will be based on clinical and biochemical data reflecting KDIGO criteria.
  Cohort 2- Chronic Kidney disease (CKD)- 20 age- and sex-matched patients with CKD will be recruited and the patients' eGFR will be matched to that of patients who had AKI and developed persistent renal impairment at the time of their interval scan (3-6 months from their baseline scan).
  Cohort 3- Control subjects- 20 age-, sex- and cardiovascular risk factor- matched control subjects will be recruited and matched to the AKI cohort.
  Cohort 4- Vasculitis- 20 patients with a new diagnosis of vasculitis (or an existing diagnosis with relapsing disease), and kidney involvement.
  Cohort 5- Kidney failure undergoing transplantation.- 20 patients with kidney failure and will receive a kidney transplant in the following 1 month.
  Cohort 6- Kidney transplant rejection- 20 patients with a biopsy proven diagnosis of transplant
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2029-11-07 (Estimated); Study Completion 2029-11-07 (Estimated)

PRIMARY OUTCOMES:
Manganese Uptake (Ki) | (baseline and follow up scan in relevant cohorts)
  Rate of manganese uptake in the kidney (cortex and medulla) and myocardium

SECONDARY OUTCOMES:
24 hour blood pressure | baseline and follow up
Arterial stiffness. | baseline and follow up
  Measure of arterial stiffness
Biomarkers of endothelial function | baseline and follow up

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised data after the end of the study will be disseminated in the public domain through the form of publications. Raw data will be retained within the study team and those researchers who will be continuing the study or further expanding the use of MEMRI will have access to this data. Anonymised data will be shared with external collaborators and scientists, subject to governance approvals.

REFERENCES:
- [Background] Legrand M, Rossignol P. Cardiovascular Consequences of Acute Kidney Injury. N Engl J Med. 2020 Jun 4;382(23):2238-2247. doi: 10.1056/NEJMra1916393. No abstract available. PMID 32492305
- [Background] Bellomo R, Kellum JA, Ronco C. Acute kidney injury. Lancet. 2012 Aug 25;380(9843):756-66. doi: 10.1016/S0140-6736(11)61454-2. Epub 2012 May 21. PMID 22617274